CLINICAL TRIAL: NCT05365867
Title: mHealth Technology to Connect and Empower People Experiencing Homelessness to Improve Health and Social Need Outcomes
Brief Title: Interactive Care Coordination and Navigation:RCT To Assess the Impact of a mHealth Intervention for Homeless Individuals
Acronym: iCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: University of Maryland (Other); Sunrise Navigation Center (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY000026665; R18HS027750 (AHRQ)
Record Dates: First submitted 2022-05-03; First posted 2022-05-09 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Number of Emergency Department and Hospital Visits Among Adults Experiencing Homelessness; Medication Adherence; Social Support; Pyschological Distress; Attainment of Social Needs (i.e., Housing, Employment, Receipt of Benefits)
Keywords: mHealth among people experiencing homelessness
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the iCAN group or usual care control group in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The biostatistician is masked to who is in the intervention or usual care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCAN Group (Experimental): iCAN is comprised of text messaging, GPS technology, preloaded apps, and telephone case management integrated within a community-based navigation center. Participants will receive 3 - 5 messages daily regarding medication adherence and appointment reminders, general health messages, motivational messages, and as needed messages for local information (e.g., weather updates). Within 48 - 72 hours of enrollment, participants will be called on their study phone by the study case manager for an intake assessment that will take 30 - 45 minutes in duration. The purpose of the assessment is to identify relevant health and social needs that the case manager can assist the participant in addressing by connecting with other medical and social services in the community. Within 48 - 72 hours of notification of a ED or hospital visit the iCAN case manager will call the participant on the study phone to assess care coordination needs for managing discharge instructions.
  Interventions: Behavioral: iCAN Group
- Usual Care Control (UCC) (No Intervention): Participants randomized to the UCC group will have access to their personal phones and use it in the usual manner with no installment of apps, text messages, or case manager interventions. Since the majority of PEH have a cell phone of some type, this will allow us to compare the intervention to how PEH typically use their cell phones. Also, the UCC will have access to all of the services available at any of the enrollment sites but no formal interaction from the iCAN case manager and no option of text messaging with the iCAN case manager.

INTERVENTIONS:
Behavioral: iCAN Group — See description in iCAN study arm.
  Arms: iCAN Group

SUMMARY:
People experiencing homelessness (PEH) are at exceptionally high risk of frequent emergency department (ED) and hospital use, poor functional outcomes, and increased morbidity and mortality from poorly managed chronic health conditions and complex social needs. Evidence-based interventions of particular promise for reducing ED and hospital utilization and improving health outcomes and meeting social needs involve:1) providing care in the community to overcome barriers including transportation and fear of stigmatization; 2) coordination of care transitions following ED or hospital discharge to improve access to needed community supports and reduce the risk of readmission; and 3) using mHealth technology to link PEH with appropriate community-based health and social services. This project builds on evidence from two feasibility studies in order to integrate and test a mHealth intervention, comprised of GPS technology and text messaging components, into a community setting to connect PEH with a community-based case manager and healthcare and social services. Our hypothesis is that integrating the mHealth intervention into an established, trusted navigation center for PEH will mitigate barriers to care and gaps in the care continuum resulting in decreased ED and hospital use and improved health outcomes and attainment of social needs. The study aim is to conduct a stratified RCT to compare a mHealth intervention with usual care community-based case management to examine the impact on healthcare utilization (primary outcome), medication adherence, social support, psychological distress and social needs attainment (secondary outcomes) in PEH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old Homeless (defined as where the person slept most nights in past 30 days (street, shelters, transitional housing, doubling-up with family or friends) Currently own a cell phone with service or use phone with wifi (when available) at baseline Currently prescribed ≥ 2 medications for chronic medical conditions (self-report) Diagnosis of at least two chronic health conditions (self-report): e.g., hypertension, diabetes, depression
* 2 hospitalizations or ED visits in the last 6 months (self-report) Score of at least 4 on the REALM-SF health literacy measure Score > 17 on the Mini-Mental State Exam

Exclusion Criteria:

Unable to communicate verbally in English. This is an exclusion criteria because the text messaging, apps, procedures and measures are not validated in in other languages.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Number of emergency department (ED) and hospital visits | Number of ED and hospital visits from baseline to 6 months post-enrollment (primary outcome), and from 6 months post-enrollment to 12 months post-enrollment (sustained impact of the intervention).
  Number of ED and hospital visits data will come from medical records from the local health information exchange.

SECONDARY OUTCOMES:
Medication Adherence | Medication adherence will be measured at baseline and 3 months and 6 months post-enrollment.
  Medication adherence will be measured using the Hill-Bone Medication Adherence Scale, a 9-item scale that measures medication adherence for chronic conditions.
Social Support | Social support will be measured at baseline and 3 months and 6 months post-enrollment.
  Social support will be measured using the modified 8-item Medical Outcomes Study Social Support Survey, a valid and reliable tool in multiple groups across various conditions.
Psychological Distress | Psychological Distress will be measured at baseline and 3 months and 6 months post-enrollment.
  The Kessler Psychological Distress Scale - 6 (K6) is comprised of 6 items that assess feelings of anxiety and depression.
Social Needs Attainment | Social need attainment will be assessed at baseline, 1, 3, 5, and 6 months post-enrollment.
  Three questions will be used to assess changes in housing and employment status and receipt of benefits.

OTHER OUTCOMES:
Process measures in iCAN group | Process measures will be collected at 1, 3, 5, and 6 months post-enrollment visits in the iCAN group.
  A number of process measures will be collected in the iCAN group. Process measures will include percentage of valid responses to text message surveys, number of case manager telephone consultations, description of type and number of case manager interventions, number of times case manager uses GPS to locate a participant, and technology issues/concerns.
Technology and Case Manager Assessment | The technology and case manager assessment will occur at the 6-month post-enrollment visit.
  At the end of the study, participants in the iCAN group will complete a modification of the Technology Acceptance Questionnaire to evaluate the acceptance of the mobile health technology and integration of case manager.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Trinity Center, Austin, Texas
  - Sunrise Navigation Center, Austin, Texas
  - Charlie Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT05365867/ICF_000.pdf